CLINICAL TRIAL: NCT02755727
Title: Platelet Rich Plasma vs Open Surgery in the Treatment of Chronic Lateral Epicondylar Tendinopathy (Tennis Elbow) A Pilot Randomized Control Trial
Brief Title: Platelet Rich Plasma vs Open Surgery in the Treatment of Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1510155
Record Dates: First submitted 2016-04-11; First posted 2016-04-29 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet Rich Plasma injection (Experimental): In the outpatient setting a sample of venous whole blood will be taken from the patient (40mls), from the antecubital fossa using standard phlebotomy techniques. The Angel™ system will be in the available also in the outpatient clinic and will be used to separate the blood to yield a PRP sample (approximately 15 minutes preparation time). The PRP sample is then injected into the common extensor origin.
  2 injections will be used per patient over 2 weeks.
  Interventions: Procedure: Platelet Rich Plasma Injection
- Open Surgical Release (Active Comparator): Standardised surgical technique based on the Nirschl technique will be used. The patient will then have a small scar centred over the lateral epicondyle and the plane opened between ECRL (Extensor Carpi Radialis Longus) and EDC (Extensor Digitorum Communis) to expose the damaged ECRB (Extensor Carpi Radialis Brevis) tendon. The amount of abnormal tendon will be documented and excised. EDC will also be inspected and any abnormal tissue documented then excised. The footprint of the excised ECRB +/- EDC is cleared of soft tissue and the bone scored with an osteotome to promote bleeding. The interval is closed with suture material and the skin wound closed.
  Interventions: Procedure: Open Surgical Release

INTERVENTIONS:
Procedure: Platelet Rich Plasma Injection — See Arms
  Arms: Platelet Rich Plasma injection
Procedure: Open Surgical Release — See arms
  Arms: Open Surgical Release

SUMMARY:
Chronic Lateral Epicondylar Tendinopathy is a debilitating condition that is associated with repetitive use of the forearm extensor muscles. Though often self-limiting in nature there are a proportion of patients who fail to respond to conservative treatments such as rest, activity modification, physiotherapy and the use of a brace. Though previously a common treatment modality steroid injections have been shown to be detrimental in the longer term. Present practice is to offer those patients who do not respond to conservative treatment surgical debridement. Though often effective this is an invasive procedure. Platelet rich plasma injections may offer a viable alternative in chronic cases however there is no systematic evidence of its efficacy.

Methods 12 patients, diagnosed with chronic lateral epicondylar tendinopathy, will be randomly assigned to receive either open surgical debridement or platelet rich plasma injections. Following treatment, they will be followed up at intervals of 6 weeks and 3, 6 and 12 months. The outcome of each treatment will be assessed using validated outcome scoring measures specifically designed for upper limb pathology. The results of this pilot study will be used to construct a larger randomised control trial.

DETAILED DESCRIPTION:
Research Question

There is no difference in patient reported outcome measures between open surgical release and platelet rich plasma injection in the treatment of chronic lateral epicondylar tendinopathy (Tennis Elbow).

Aims

* To estimate the distribution of patient-reported outcome measures (PROMS) at 6 weeks, 3 months, 6 months and 1 year
* To record any adverse events associated with either treatment
* To test the feasibility of the study design in preparation for a larger randomised trial
* To collect data that will allow a power calculation for a larger randomised trial
* To use the data for a larger grant application

Objectives

* To randomise patients who have failed conservative management of tennis elbow to one of two treatment methods: Platelet Rich Plasma or Open Surgical Release
* To collect treatment outcome data in the form of a visual analogue scale, Oxford Elbow Score and DASH (Disability of Arm, Shoulder and Hand) score
* To use the current best guidance and administer leucocyte-rich PRP (L-PRP) under ultrasound guidance
* To use the data gained from a pilot study to assess the viability of a larger randomised control trial

Research design This pilot study will be conducted as a randomised controlled pilot trial at the Royal Devon and Exeter Hospital, UK.

Patient Selection Patients will be selected from those who attend the outpatient elbow clinic at the Royal Devon and Exeter Hospital. All patients will be reviewed by a Consultant Orthopaedic Surgeon specialised in Elbow surgery. The inclusion criteria will be any patient who has experienced more than 6 months of symptoms from tennis elbow, that include pain on the lateral elbow that radiates down the forearm, point tenderness over the origin of the extensor muscles or at its close proximity (within 2.5cm) and pain on resisted extension of the Wrist. Patients must also have failed conservative treatment (a course of physiotherapy and activity modification) and have a baseline elbow pain >3/10 on VAS during resisted elbow extension.

Patients will be excluded: in the presence of a full tendon tear on pre-intervention ultrasound, are unfit for surgical intervention, have undergone previous elbow surgery, have previously undergone PRP injection therapy, systemic autoimmune rheumatological disease, receiving immunosuppressive treatments, received local steroid injection within 3 months of randomization or are unable to comply with follow-up.

Intervention The 2 arms of the trial will include PRP therapy or Open surgical debridement

* Platelet Rich Plasma injection
* Open Surgical Release (presently standard treatment regimen)

Both groups of patients will be given an identical physiotherapy programme and followed-up at identical timeframes to record the outcomes of the interventions.

Sample size The present proposal is intended to be a pilot study. As such the intention will be to randomise 6 patients to each arm of the trial, 12 patients in total. It has been estimated that 1 suitable patient is likely to be seen in the outpatient clinic each week. Owing for attrition and patient suitability it is hoped that a 6 month enrolment period will yield 12 patients.

Randomisation The participating patients will be randomised in a 1:1 allocation to open surgery or PRP injections. The randomisation will be administered by a central independent randomisation service, provided by a medical secretary using a computer-generated randomisation sequence and sealed in sequentially numbered envelopes, who is completely independent of the trial.

Outcome scoring Primary outcome measures will be in the form of Patient Reported Outcome Measures (PROMS) and Range of Motion (ROM) Primary Outcome: Change in Patient Rated Tennis Elbow Evaluation (PRTEE) between pre-intervention and at 3 months post-intervention - patient compiled questionnaire based on specific elbow symptoms of Tennis Elbow

All secondary outcome measures to be completed pre-operatively and at 6 weeks, 3 months, 6 months and 12 months.

● PROMS Visual Analogue Scale (VAS) - Using a linear scale of 10cms length. Assessed through change in score over time.

Disabilities of the Arm, Shoulder and Hand (quickDASH) - patient compiled questionnaire based on subjective assessment of symptoms and abilities to perform activities of daily living over the last week.

Oxford Elbow Score (OES) - patient compiled questionnaire based on specific elbow symptoms related activities of daily living over the past 4 weeks.

Adverse events - peri-procedural, 6 weeks, 3 months, 6 months and 12 months

ELIGIBILITY:
Inclusion Criteria:

Any patient who:

* Has experienced more than 6 months of symptoms from tennis elbow (pain on the lateral elbow that radiates down the forearm, point tenderness over the origin of the extensor muscles or at its close proximity (within 2.5cm) and pain on resisted extension of the Wrist).
* Patients must also have failed conservative treatment (a course of physiotherapy and activity modification)
* Baseline elbow pain >3/10 on VAS during resisted elbow extension.

Exclusion Criteria:

* Presence of a full tendon tear on pre-intervention ultrasound
* Unfit for surgical intervention
* Have undergone previous elbow surgery,
* Have previously undergone PRP injection therapy
* Systemic autoimmune rheumatological disease
* Receiving immunosuppressive treatments
* Received local steroid injection within 3 months of randomization
* Unable to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Patient Rated Tennis Elbow Evaluation (PRTEE) | To be completed pre-intervention and at 3 months post-intervention
  patient compiled questionnaire based on specific elbow symptoms of Tennis Elbow

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) | To be completed pre-operatively and at 6 weeks, 3 months, 6 month and 12 months post-intervention
  - Using a linear scale of 10cms length. Assessed through change in score over time.
Change in Disabilities of the Arm, Shoulder and Hand (quickDASH) | To be completed pre-operatively and at 6 weeks, 3 months, 6 month and 12 months post-intervention
  - patient compiled questionnaire based on subjective assessment of symptoms and abilities to perform activities of daily living over the last week.
Change in Oxford Elbow Score (OES) | To be completed pre-operatively and at 6 weeks, 3 months, 6 month and 12 months post-intervention
  - patient compiled questionnaire based on specific elbow symptoms related activities of daily living over the past 4 weeks.
Adverse events | peri-procedural, 6 weeks, 3 months, 6 months and 12 months
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: C Gardener, Study Chair — Research Development Directorate - Royal Devon and Exeter Hospital
Locations (1):
- Royal Deveon and Exeter Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No